CLINICAL TRIAL: NCT05697562
Title: A Randomized Comparative Evaluation of Superior Rectal Arterial Embolization in Hemorrhoidal Disease
Brief Title: Evaluation of Superior Rectal Arterial Embolization in Hemorrhoidal Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEMbol
Record Dates: First submitted 2022-12-21; First posted 2023-01-26 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Intervention Model Description: Patients will be divided in 2 groups: Anticoagulation group (A) and No Anticoagulation group (NA), based on their regular medication. In both groups, A and NA, are 2 study arms, resp. DG HAL as standard clinical practice versus SRAE (group A) and RBL as standard clinical practice versus SRAE (arm NA). See figure below.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- anticoagulation group with DG HAL (Placebo Comparator)
  Interventions: Procedure: Doppler-Guided Hemorrhoidal Artery Ligation (DG-HAL)
- anticoagulation group with SRAE (Active Comparator)
  Interventions: Procedure: Superior Rectal Artery Embolization (SRAE)
- no anticoagulation group with RBL (Placebo Comparator)
  Interventions: Procedure: Rubber band ligatures (RBL)
- no anticoagulation group with SRAE (Active Comparator)
  Interventions: Procedure: Superior Rectal Artery Embolization (SRAE)

INTERVENTIONS:
Procedure: Rubber band ligatures (RBL) — This instrumental technique is realized during consultation. A rubber band is applied on top of each hemorrhoidal complex via a proctoscope. This banding causes an ulceration which heals with resulting fibrosis. The patient can receive a maximum of 3 RBL during each session, which can be repeated up to 3 times at a 6 weeks interval.
  Arms: no anticoagulation group with RBL
Procedure: Superior Rectal Artery Embolization (SRAE) — This technique is realized under local anesthesia during a one-day hospitalization. The interventional radiologist will perform the procedure in the angiography room. After local anesthesia right femoral artery puncture is performed and a 4 F or 5 F introducer sheath is placed using the Seldinger technique. With an appropriate 4 or 5 F catheter the superior rectal artery is catheterized. With a microcatheter the different branches are selectively occluded with microcoils. The endpoint of embolization is reached when all SRA branches above the pubic ramus are embolized, with cessation of flow distally or a static column of contrast.
  The procedure can be repeated with addition of the embolization of the middle rectal wall artery (MRA) in case of failure after 12 weeks.
  Arms: anticoagulation group with SRAE; no anticoagulation group with SRAE
Procedure: Doppler-Guided Hemorrhoidal Artery Ligation (DG-HAL) — The procedure is performed in lithotomy position with a modified proctoscope including a Doppler transducer (THD device) under anesthesia during a one-day hospitalization. This transanal Doppler guidance enables accurate detection and targeted suture ligation of the SRAs Following gel lubrication, the proctoscope is inserted through the anal canal reaching the low rectum, about 6-7 cm from the anal verge. After identification of the best place for artery ligation, the Doppler system is turned off. The artery will be directly ligated with a Z-stitch at the site of the best Doppler signal.
  Arms: anticoagulation group with DG HAL

SUMMARY:
SRAE is a promising treatment of bleeding HD as a minimally invasive approach without sphincter damage nor direct mucosal anorectal trauma. Feasibility, efficacy and safety were studied in several trials. A randomized controlled study should confirm the benefits of this technique and will define its therapeutic role in HD.

Embolization and DG-HAL are based on the same concept of vascular occlusion of hemorrhoidal branches of the rectal artery. Furthermore, DG-HAL and RBL are equally effective procedures. The assumption is that treatment with SRAE is not inferior in comparison to RBL or DG HAL in respectively patients without or with antiplatelet/anticoagulation therapy in terms of symptom control and bleeding (non-inferiority study).

DETAILED DESCRIPTION:
Hemorrhoidal disease (HD) is the most common anorectal pathology. Therapeutic management of HD ranges from conservative treatment and instrumental treatment to surgical approach. Beside these, certain minimally invasive techniques such as radiofrequency ablation, laser coagulation and Superior Rectal Artery Embolization (SRAE) are gaining interest. SRAE is a promising treatment of bleeding HD as a minimally invasive approach without sphincter damage nor direct mucosal anorectal trauma. Feasibility, efficacy and safety were studied in several trials. A randomized controlled study should confirm the benefits of this technique and will define its therapeutic role in HD. Embolization and DG-HAL are based on the same concept of vascular occlusion of hemorrhoidal branches of the rectal artery. Furthermore, DG-HAL and RBL are equally effective procedures. The assumption is that treatment with SRAE is not inferior in comparison to RBL or DG HAL in respectively patients without or with antiplatelet/anticoagulation therapy in terms of symptom control and bleeding (non-inferiority study).

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for Hemorrhoidal disease with bleeding are eligible. Significant bleeding is defined as a HBS of ≥ 5.
* Age > 18 years old;
* Sexes eligible for study: all
* Hemorrhoidal disease grade I-III according the Goligher classification with rectal bleeding as predominant symptom
* History of prior instrumental treatment of HD does not prohibit inclusion
* Able to understand and read Dutch, French or English

Exclusion Criteria:

* Permanent hemorrhoidal prolapse/grade IV hemorrhoidal disease
* Rectal prolapse
* History of proctological surgery for HD
* Acute complicated course of HD i.e. acute thrombosis (fluxio hemorrhoidalis or perianal hematoma)
* Anal stenosis, congenital of acquired
* Chronic anal fissure
* Active rectal inflammation, including peri-anal abscess (e.g. Inflammatory Bowel Disease, infectious,…)
* History of colorectal or anal cancer
* History of rectal or sigmoidal resection
* Portal hypertension and liver cirrhosis Child Pugh C
* Radiation rectitis
* Neurological disease involving anal sphincter musculature
* Severe psychiatric disorder
* Pregnancy
* Allergy to iodinated contrast agents
* Colorectal neoplasia as the cause of bleeding (excluded with a (virtual) colonoscopy in the last year)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
symptom control | from baseline to 3 months
  the main objective is to control the symptoms, for this the Hemorrhoidal Bleeding Score is to be used

SECONDARY OUTCOMES:
Symptom control | from baseline to 12 months
  a secondary objective is to control the symptoms, for this the Hemorrhoidal Bleeding Score is to be used
Patient reported effectiveness | from baseline till 12 months
  a secondary objective is to report patient effectiveness, this will be measured using Patient-Reported Outcome Measure-Haemorrhoidal Impact and Satisfaction score (PROM-HISS)
Patient reported effectiveness | from baseline till 12 months
  a secondary objective is to report patient effectiveness, this will be measured using the 5-level EQ-5D-5L score
clinical effectiveness | from baseline till 12 months
  a secondary objective is to report clinical effectiveness, this will be measured using the Goligher score
prevalence of complications | from baseline till 12 months
  a secondary objective is to report the prevalence of complications, this will be measured using among others the pain score reported by Visual Analogue Scale (VAS)
prevalence of re-interventions | from baseline till 12 months
  a secondary objective is to report the prevalence of re-interventions, this will be measured among others with the pain score reported by Visual Analogue Scale (VAS)
prevalence of fecal incontinence | from baseline till 12 months
  a secondary objective is to report the prevalence of fecal incontinence, this will be measured using the Jorge-wexner score

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Belgium

IPD SHARING:
Plan to Share IPD: No